CLINICAL TRIAL: NCT06209970
Title: Injection of 35kDa Hyaluronan Fragment Alleviates Pain Associated With Radiotherapy for Treatment of Colorectal and Rectal Cancer
Brief Title: 35kDa Hyaluronan Fragment Treatment of Colorectal and Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20231218
Record Dates: First submitted 2023-12-18; First posted 2024-01-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-12

CONDITIONS: Cancer Pain
Keywords: 35kDa hyaluronan fragment; pain; colorectal cancer; rectal cancer
MeSH Terms: conditions — Cancer Pain; Pain; Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35kDa hyaluronan fragment HA35 injection (Experimental): A total of 2000 units of bovine testis hyaluronidase PH20 (hyaluronidase for injection H31022111, P.R.C) and 100 mg high molecular weight HA (sodium hyaluronate for injection, H20174089, P.R.C) were mixed at room temperature for 20 minutes, then was locally injected into patient's abdominal deep fat layer by a registered nurse or a physician in order to quickly alleviate pain associated with radiotherapy for treatment colorectal and rectal cancer.
  Interventions: Drug: HA35

INTERVENTIONS:
Drug: HA35 — All the freshly made HA35 or B-HA samples were diluted to a final concentration of 5 mg/ml. The filter membrane with 220nm pore size was used to filter freshly made HA35 or B-HA injection in order to test its human tissue permeability as <220nm nino-particle.

SUMMARY:
HA35 (Bioactive HA or B-HA or HA35) have good tissue permeability (B-HA injection, Ministry of Health, Registration number L20200708MP07707). HA35 might not lose HA's bioactivities of binding to a variety of hyaluronan's binding proteins or receptors, including the analgesic and anticancer effects of hyaluronan, therefore being named bioactive HA or B-HA (10) (B-HA injection, Ministry of Health, Registration number L20200708MP07707).

DETAILED DESCRIPTION:
The previous study has shown that naked mole rat who has high tissue content of hyaluronan and its fragments is insensitive to pain. The previous study has also shown that hyaluronan modulates pain-regulated TRPV1 channel opening, reducing peripheral nociceptor activity and pain. The previous study has again shown that local injection of 35kDa hyaluronan fragment HA35 is effective in treating inflammatory and neuropathic pain. This study employs freshly made HA35 injection for treatment of pain associated with radiotherapy for treatment of colorectal and rectal cancer. A numerical rating scale from 0 to 10 was used to assess the pain after 1 hour, 3 hours, 24 hours, 48 hours and 72 hours of the injection.

ELIGIBILITY:
Inclusion Criteria:

* All patients had different degrees of metastasis of the cancers, including bone metastasis.
* All patients undergo targeted radiotherapy shortly before this study.
* All the patient volunteers included in this study were allowed to use antibiotic compounds on and off during the treatment in order to prevent possible infection associated with the cancers for ethnic consideration.
* The included patients were aged 48 to 60 years.

Exclusion Criteria:

* Can not independently determine the level of pain.
* Severe bleeding and severe inflammation

Ages: 48 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 1 hour, 3 hours, 24 hours, 48 hours and 72 hours
  A numerical rating scale (NRS) from 0 to 10 was used to assess the pain after 1 hour, 3 hours, 24 hours, 48 hours and 72 hours of the injection. Each patient rates their pain on a scale of 0 to 10, where a score of 0 means "no pain" and 10 means "the most painful". More specifically, 0 points indicates no pain; 1-3 points can be interpreted as slight and bearable pain; 4-6 points can be interpreted as pain that affects sleep but is still tolerable; and 7-10 points can be interpreted as intense and unbearable pain that affects sleep or other activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Huinorde Science and Technology Co.,Ltd, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No